CLINICAL TRIAL: NCT02471898
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Four-Part Evaluation of the Efficacy and Safety of Locally Administered HTX-011 for Postoperative Analgesia Following Bunionectomy
Brief Title: A Phase 2, Two-Part Evaluation of the Efficacy and Safety of Locally Administered HTX-011 for Postoperative Analgesia Following Bunionectomy
Acronym: HTX-011
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTX-011-C2015-201
Record Dates: First submitted 2015-06-09; First posted 2015-06-15 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HTX-011 (Experimental): Evaluate the analgesic efficacy of HTX-011
  Interventions: Drug: HTX-011
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTX-011
  Arms: HTX-011
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Two-Part Evaluation of the Efficacy and Safety of Locally Administered HTX-011 for Postoperative Analgesia Following Bunionectomy

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent.
2. Male or female between 18 and 65 years of age, inclusive.
3. Be scheduled to undergo a primary unilateral first metatarsal bunionectomy repair, without collateral procedures, under regional anesthesia
4. Be American Society of Anesthesiology (ASA) physical Class 1 or 2.
5. Female subjects are eligible only if all of the following apply:

   * Not pregnant (female subject of child bearing potential must have a negative serum pregnancy tests at screening and negative urine pregnancy test before surgery);
   * Not lactating
   * Not planning to become pregnant during the study
   * Be surgically sterile; or at least two years post-menopausal; or have a monogamous partner who is surgically sterile; or is practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening visits and commits to the use of an acceptable form of birth control for the duration of the study and for 30 days from completion of the study.
6. Male patients must be surgically sterile (biologically or surgically) or commit to the use of a reliable method of birth control for the duration of the study until at least 1 week after the administration of study medication.
7. Have a body mass index ≤ 35 kg/m2.
8. Be able to understand the study procedures, comply with all study procedures, and agree to participate in the study program.
9. Be able to understand and communicate in English.

Exclusion Criteria:

1. Have a known allergy to Bupivacaine/Meloxicam or any HTX-011/placebo excipient or to any peri- or postoperative medications used in this study including oxycodone lidocaine, propofol, fentanyl, and midazolam.
2. Have a clinically significant abnormal clinical laboratory test value according to the judgment of the investigator.
3. Have history of or positive test results for HIV or hepatitis B or C at screening.
4. Have, as determined by the investigator or the study's medical monitor, a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study.
5. Have a history of migraine or frequent headaches, seizures, or are currently taking anticonvulsants.
6. Have another painful physical condition that, in the opinion of the investigator, may confound the assessments of postoperative pain.
7. Have been receiving or have received chronic opioid therapy defined as greater than 15 morphine equivalents units per day for greater than 3 out of 7 days per week over a one-month period within 12 months of study treatment initiation.
8. Use concurrent therapy that could interfere with the evaluation of efficacy or safety, such as any drugs which in the investigator's opinion may exert significant analgesic properties or act synergistically with HTX-011-19.
9. Have evidence of a clinically significant 12-lead ECG abnormality according to the judgment of the investigator.
10. Have a history of alcohol abuse (regularly drinks > 4 units of alcohol per day; 8 oz. beer, 3 oz. wine, 1 oz. spirits) or prescription/illicit drug abuse.
11. Have positive results on the alcohol breath test indicative of alcohol abuse or urine drug screen indicative of illicit drug use (unless results can be explained by a current prescription or acceptable over-the-counter medication at screening as determined by the investigator; however, the urine drug screen at prior to surgery must be negative) at screening, and/or prior to surgery.
12. Unable to discontinue medications that have not been at a stable dose for at least 14 days prior to the scheduled bunionectomy procedure, within 5 half-lives of the specific prior medication (or, if half-life is not known, within 48 hours) before dosing with study medication.
13. Have utilized corticosteroids, either systemically, inhaled either intranasally or orally, or by intra-articular injection, within 14 days prior to the study surgical procedure.
14. Have received any investigational product within 30 days before dosing with study medication.
15. Have previously received HTX-011-19 in clinical trials or had bunionectomy in the last 3 months.
16. Experiences a clinically significant event during surgery prior to the administration of the investigational product (e.g., excessive bleeding, hemodynamic instability) that would render the subject medically unstable, complicate their postsurgical course, or significantly increase the risk of study drug administration as per the judgment of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
SPI0-24 | 24 hours
  Summed Pain Intensity Scores over the first 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Pasadena, California, United States